CLINICAL TRIAL: NCT01652404
Title: PROcalcitonin to SHORTen Antibiotics Duration in PEDiatricICU Patients (ProShort-Ped) Trial
Acronym: ProShort-Ped
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Children's Hospital (Other Government)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN01
Record Dates: First submitted 2011-08-22; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Sepsis
Keywords: ICU; sepsis; antibiotic therapy; procalcitonin
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Procalcitonin-guided treatment (Experimental): The duration of antibiotics will be determined by the procalcitonin levels.
  Interventions: Behavioral: Procalcitonin-guided treatment
- Conventional treatment (Active Comparator): The duration of antibiotics will be determined by the treating physician.
  Interventions: Behavioral: Conventional treatment

INTERVENTIONS:
Behavioral: Procalcitonin-guided treatment — The antibiotics duration will be determined by the serum procalcitonin level at day 5, 7 and 9.
  Arms: Procalcitonin-guided treatment
Behavioral: Conventional treatment — The antibiotics duration will be determined by treating physician.
  Arms: Conventional treatment

SUMMARY:
The purpose of this study is to give conclusive evidence on whether serial PCT (Procalcitonin) measurements can facilitate individual decision-making and shorten antibiotic treatment duration in patients with sepsis in the pediatric ICU (Intensive Care Unit).

DETAILED DESCRIPTION:
In this study, the investigators aimed to design a multi-center trial addressing aforementioned flaws. The investigators will set stricter inclusion criteria, collect complete data on relapse or secondary infection, and include sufficient number of patients to show non-inferiority to conventional therapy by a delta margin of 10% [11]. The investigators aimed to give conclusive evidence on whether serial PCT measurements can facilitate individual decision-making and shorten antibiotic treatment duration in patients with sepsis in the pediatric ICU.

ELIGIBILITY:
Inclusion Criteria:

All patients with laboratory- or image-confirmed severe infection at admission or during stay in pediatric ICU will be eligible for inclusion.

* Definition of laboratory- or image-confirmed severe infection:

* Two or more of four signs of inflammation:

  * Temperature >38.3℃ or <36℃
  * Heart rate > 90 beats/min
  * Respiratory rate >20 breaths/min or PaCO2 (Arterial pressure of carbon dioxide) < 32 mmHg
  * WBC (White Blood Cell count) > 12,000 cells/mm3, <4000 cells/mm3, or >5% band-form WBC
* Initial Procalcitonin > 0.5 ng/mL
* Presence of either laboratory or image evidence of infection
* Laboratory evidence: Sign of inflammation in urine, CSF (Cerebrospinal Fluid), ascites, pleural effusion or local abscess
* Image evidence: Compatible findings on Chest X ray, ultrasound, CT (Computed Tomography), MR image (Magnetic Resonance Image)

Exclusion Criteria:

* Age greater than 15 years or less than 1 month
* Known pregnancy
* Expected ICU stay less than 3 days
* Neutropenia: ANC (Absolute Neutrophil Count) <500/mm3
* Specific infections for which long-term antibiotic treatment is strongly recommended:

  * Lobar pneumonia or empyema
  * Bacterial meningitis
  * Osteomyelitis
  * Infective endocarditis
  * Local abscess
  * Mediastinitin

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Average antibiotics duration | 28 days
  Efficacy endpoint
28-day mortality rate | 28 days
  Safety endpoint

SECONDARY OUTCOMES:
Proportion of antibiotics use in both arms | 28 days
  Efficacy endpoint
Length of ICU stay | 90 days
  Efficacy endpoint
Recurrence of fever within 72 hours of antibiotics discontinuation | 28 days
  Safety endpoint
SOFA score (Sequential Organ Failure Assessment score) | 28 days
  Safety endpoint
Reinfection rate between 72-hours and 28 days post antibiotics discontinuation | 28 days
  Safety endpoint
90-day all-cause mortality | 90 days
  Safety endpoint
90-day readmission rate | 90 days
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Lee, MD, MSc, Principal Investigator — National Taiwan University Hospital; Yi-Min Zhu, BSc, Study Chair — Hunan Children's Hospital
Locations (1):
- Hunan Children's Hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Michael M, Hodson EM, Craig JC, Martin S, Moyer VA. Short versus standard duration oral antibiotic therapy for acute urinary tract infection in children. Cochrane Database Syst Rev. 2003;(1):CD003966. doi: 10.1002/14651858.CD003966. PMID 12535494
- [Background] Lee SL, Islam S, Cassidy LD, Abdullah F, Arca MJ; 2010 American Pediatric Surgical Association Outcomes and Clinical Trials Committee. Antibiotics and appendicitis in the pediatric population: an American Pediatric Surgical Association Outcomes and Clinical Trials Committee systematic review. J Pediatr Surg. 2010 Nov;45(11):2181-5. doi: 10.1016/j.jpedsurg.2010.06.038. PMID 21034941